CLINICAL TRIAL: NCT04613362
Title: TENACITY: TelemEdiciNe-bAsed Cognitive Therapy for Migraine
Brief Title: TelemEdiciNe-bAsed Cognitive TherapY for Migraines
Acronym: TENACITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRP 20-002
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Migraine Headache
Keywords: Implementation Science; Telehealth; Cognitive Behavioral Therapy
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled feasibility pilot with a single intervention arm, and a usual care control arm. The intervention arm includes participation in the TENACITY telehealth cognitive behavioral therapy CBT program for headache plus education. The usual care arm includes behavioral treatment as usual which may include outpatient clinic-based health psychology in the VA or in the community, or mindfulness sessions by LCSW.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be randomized by mode of delivery to the telehealth or TAU treatment stratified by site (VA Medical Center). Upon completion of the baseline evaluation, the project coordinator will assign random assignment. The research assistants will be masked to random assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TENACITY Telehealth Cognitive Behavioral Therapy for Migraine (Experimental): Six sessions of standardized Cognitive Behavioral Therapy for patients with diagnosed chronic migraine headaches will be delivered by a clinical health psychologist via telehealth platform. All patients have access to a set of standardized educational, headache self-management materials.
  Interventions: Behavioral: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine
- Behavioral Usual Care (Active Comparator): Behavioral usual care may include outpatient clinic-based health psychology in the VA or Community Care, or mindfulness sessions with LCSW. Behavioral usual care will be delivered by clinicians for patients with diagnosed chronic migraine.
  Interventions: Behavioral: Behavioral Usual Care

INTERVENTIONS:
Behavioral: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine — Clinical health psychology therapy delivered via telehealth
  Arms: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine
Behavioral: Behavioral Usual Care — Behavioral usual care may include outpatient clinic-based health psychology in the VA or Community Care, or mindfulness sessions with LCSW.
  Arms: Behavioral Usual Care

SUMMARY:
The goal of this pilot study is to evaluate a bundle of implementation strategies at three Veteran Affairs Medical Centers (VAMCs) to facilitate the referral and adoption of a telehealth based, cognitive behavioral therapy program delivered by Health Psychologists for Veterans with chronic migraine to inform a future fully-powered hybrid type 2 effectiveness-implementation design. Veteran patients will be randomized to either the telehealth delivered CBT or usual care. Headache symptoms and severity will be reported using a VA text messaging application.

DETAILED DESCRIPTION:
With VHA's infrastructure dedicated to efficient telehealth delivery into patient homes, the delivery of a behavioral intervention for chronic migraine, CM, via the telehealth platform is primed to address barriers of in-person care delivery and holds considerable promise to reach and improve Veteran headache-related quality of life. Therefore, the goal is to evaluate an adapted bundle of EB implementation strategies to increase adoption of a Telemedicine-based Cognitive Behavioral Therapy (CBT) program (TENACITY) for CM in 2 VA HCoEs (VA Connecticut Healthcare System [VACHS], a large, multi-disciplinary HCoE, and Birmingham VA Medical Center [BVAMC], a smaller VA Headache Consortium Center. The HCoEs are charged with improving headache care throughout the VA, not just within an individual VAMC. As part of this study, a non-HCoE will also participate, providing an opportunity for the TENACITY study to extend this virtual specialty headache care to Veterans without headache specialty care. Dallas VA Medical Center, also known as the North Texas Health Care System [NTHCS] will participate as a third site.

The investigators will determine whether TENACITY can be efficiently delivered through the vehicle of telehealth by conducting a pilot randomly controlled trial (RCT) comparing a) TENACITY to b) behavioral treatment as usual (TAU; i.e., behavioral usual care).

The investigators will recruit Veterans diagnosed with chronic migraine during the one-year recruitment period across the 3 VAMCs. The investigators will randomize eligible Veterans to participate either in the TENACITY intervention (n=50) or treatment as usual (n=50).

The specific aims are threefold:

Aim 1: To develop a bundle of evidence-based practice (EBP) implementation strategies to engage 3 VA Medical Centers [2 Headache Centers of Excellence HCoEs and 1 general neurology service] and facilitate their local adaptation and implementation of Cognitive Behavioral Therapy (CBT) (TENACITY) through the vehicle of telehealth services.

Aim 2. To conduct a pilot RCT and determine the preliminary efficacy and feasibility of TENACITY compared to TAU across 3 VA sites.

Hypothesis 2: Veterans receiving TENACITY will experience a statistically significant reduction in routine clinical headache metrics: headache frequency [headache days per month] (primary outcome), headache-related impairment and psychological symptoms (secondary outcomes) compared to usual care at 3 and 6 months.

Aim 3: The investigators will conduct exploratory cost analysis of TENACITY from the Veteran's perspective, using inputs from the pilot RCT, and a two-year budget impact analysis from the VHA's perspective, incorporating the costs of implementation as well as direct costs (and cost-savings,) of providing the TENACITY intervention over all HCoEs to VHA.

Hypothesis 3: TENACITY will be cost-effective and provide value to Veterans and VHA.

ELIGIBILITY:
Inclusion Criteria:

Veteran patients eligible to participate must have:

* A chronic migraine headache ICD-10 diagnosis;
* Completion of at least 28 headache diary days;
* A confirmed frequency of at least 8 headache days per month;
* A primary complaint of headache

Exclusion Criteria:

Veteran patients not eligible to participate include:

* Non-Veterans;
* Veteran patients without a CM headache ICD-10 diagnosis;
* Veteran patients whose primary pain complaint is not headache;
* Veteran patients who have received greater than or equal to 90 days of opioid therapy for chronic low back pain from the date of chart screening;
* Veteran patients who do not speak English;
* Veteran patients who have a current diagnosis of severe cognitive impairment indicated by clinical provider, medical chart, or Short Portable Mental Status Questionnaire (SPMSQ);
* Veteran patients who have Post Traumatic headache;
* Veteran patients who have a diagnosis of cluster headache, other primary headache, post-whiplash headache, secondary headache, or trigeminal autonomic cephalalgia.
* Any patients currently suffering from a disabling psychiatric illness (as noted by clinician);
* Veteran patients who self-report Traumatic Brain Injury less than or equal to 1 year before diagnosis of Chronic Migraine, or worsening of Chronic Migraine.
* Veteran patients who relate daily suicidal ideation within the last 2 weeks as indicated by the PHQ-9 with an answer of "3" to question nine;
* Veteran patients who have severe depression, as indicated by PHQ-9 score greater than or equal to 20;
* Veteran patients who are deemed by clinicians who are unable to participate in this trial;
* Patients who are terminally ill (life expectancy of <12 months as noted by clinician);
* Patients who are homeless or live in long-term care, nursing home, rehabilitation, or domiciliary services, etc.
* Veteran patients who decline to or cannot use the Annie App;
* Veteran patients who decline to or cannot use My HealtheVet secure messaging
* Veteran patients who have been treated by a HCoE clinical health psychologist in the last two years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M. Damush, PhD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (4):
- United States (4):
  - Birmingham VA Medical Center, Birmingham, AL, Birmingham, Alabama
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
After the study completion and the planned and secondary analyses are published by the study team, a limited de-identified data set will be made available upon request for a limited period.
Time Frame: To be determined

REFERENCES:
- [Result] Goldman RE, Damush TM, Kuruvilla DE, Lindsey H, Baird S, Riley S, Burrone Bs L, Grinberg AS, Seng EK, Fenton BT, Sico JJ. Essential components of care in a multidisciplinary headache center: Perspectives from headache neurology specialists. Headache. 2022 Mar;62(3):306-318. doi: 10.1111/head.14277. Epub 2022 Mar 16. PMID 35293614
- [Result] Seng EK, Fenton BT, Wang K, Lipton RB, Ney J, Damush T, Grinberg AS, Skanderson M, Sico JJ. Frequency, Demographics, Comorbidities, and Health Care Utilization by Veterans With Migraine: A VA Nationwide Cohort Study. Neurology. 2022 Oct 31;99(18):e1979-e1992. doi: 10.1212/WNL.0000000000200888. PMID 36100439

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on physician referral and recruitment cohort lists at 3 VA medical centers between April 2021 and April 2022. The first participant was enrolled on April 22, 2021 and the last participant was enrolled on April 29, 2022. All study procedures were conducted virtually and via telephone.
Pre-assignment Details: Of 80 enrolled participants, 57 met inclusion criteria after an initial screening phase and were randomized to treatment. Exclusions were as follows: less than 28 headache diary days completed (n=13), less than 8 headache days per month (n=7), and lost to follow-up (n=3).
Period: Intervention Period
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Started | 30 | 27
Received Intervention | 27 | 17
Did Not Receive Intervention | 3 | 10
Completed | 30 | 27
Not Completed | 0 | 0
Period: 3 Month Follow-up
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Started | 30 | 27
Completed | 29 | 25
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2
Period: 6 Month Follow-up
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Started | 29 | 25
Completed | 29 | 24
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Veteran patients with a migraine headache diagnosis receiving care in the Veterans Healthcare Administration and had confirmed chronic headache through a headache diary.
Groups:
- Total: Total of all reporting groups
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care | Total
Number analyzed (Participants) | 30 | 27 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 26 | 55
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 5 | 16
  White | 14 | 17 | 31
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Headache Days at 3 Months
Description: Daily self-reported migraine headaches using a VA text message protocol
Time Frame: 3 Months after Baseline
Measure: Mean (Standard Deviation); unit: headache days
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 30 | 27
headache days
  Baseline | 18.17 (7.82) | 19.19 (8.54)
  3 months | 16.47 (10.17) | 18.26 (11.05)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; Test type: Superiority; p = 0.61, Mixed Models Analysis — adjusted for gender which is included as a covariate; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.34 to 1.97]

2. Primary Outcome: Budget Impact Analysis - Cost of Training (Implementation)
Description: Costs associated with program implementation
Time Frame: 2 years
Population: Summary Costs
Measure: Number; unit: dollars
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 30 | 27
dollars | 12020.99 | 271.57

3. Other Pre Specified Outcome: Migraine-Specific Quality of Life Questionnaire (MSQ)
Description: The MSQ is a 14-item measure of headache-related quality of life. Higher scores indicate a higher quality of life. Unscaled scores range from 0 to 70.
Time Frame: 3 months, 6 months
Population: The number analyzed in one or more rows differs from overall number analyzed because some participants chose to not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 24 | 24
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 48.39 (23.07) | 57.06 (19.36)
  6 months: number analyzed (Participants) | 24 | 22
  6 months | 48.79 (24.29) | 53.32 (16.72)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 month; Test type: Superiority; p = 0.1724, Mixed Models Analysis; Mean Difference (Net) = -8.8028, 95% CI 2-sided [-21.5314 to 3.9257], Standard Error of Mean 6.3895
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.4399, Mixed Models Analysis; Mean Difference (Net) = -4.6533, 95% CI 2-sided [-16.5917 to 7.2851], Standard Error of Mean 5.9929

4. Other Pre Specified Outcome: Migraine Disability Assessment (MIDAS)
Description: The MIDAS is a 5-item, self-report measure of disability related to headache based on number of missed or significantly limited activity days due to headache in school or paid work, household work, and family, social, or leisure activities. Responses are categorized as follows: little or no disability (0-5), mild disability (6-10), moderate disability (11-20), and severe disability (21+). Scale has a range from 0 to 270, with a higher score indicating a worse outcome.
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 23 | 22
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 83.09 (68.72) | 64.94 (47.59)
  6 months | 63.17 (61.88) | 68.68 (61.40)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.3021, Mixed Models Analysis; Mean Difference (Net) = 18.7886, 95% CI 2-sided [-17.2261 to 54.8032], Standard Error of Mean 18.0826
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.7624, Mixed Models Analysis; Mean Difference (Net) = -5.1996, 95% CI 2-sided [-39.3245 to 28.9254], Standard Error of Mean 17.1338

5. Other Pre Specified Outcome: Headache-specific Pain Catastrophizing Scale (HPCS)
Description: The HPCS is a modified version of the validated Pain Catastrophizing Scale (substitutes "headache" for "pain" in the questions). The HPCS is a 13-item measure used to assess catastrophic thinking related to headache. Item responses range from 0 to 4 (0 = not at all, 4 = all the time). Total scores range from 0 to 52, with higher scores indicating higher levels of catastrophizing.
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 23 | 22
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 26.69 (17.05) | 20.88 (9.69)
  6 months | 23.55 (18.57) | 23.84 (11.66)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.1783, Mixed Models Analysis; Mean Difference (Net) = 5.9613, 95% CI 2-sided [-2.7794 to 14.7019], Standard Error of Mean 4.3867
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.959, Mixed Models Analysis; Mean Difference (Net) = -0.2145, 95% CI 2-sided [-8.4965 to 8.0675], Standard Error of Mean 4.1565

6. Other Pre Specified Outcome: Headache Management Self-Efficacy Scale (HMSE)
Description: The HMSE is a 25-item measure used to assess a participant's perception of their ability to take actions to prevent and manage their headaches and headache-related disability. Item responses range from 1 to 7 (1 = strongly disagree, 7 = strongly agree). Total scores range from 25 to 175 with higher scores indicating higher levels of headache management self-efficacy.
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 24 | 22
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 101.09 (26.16) | 113.39 (19.37)
  6 months | 103.97 (31.04) | 111.00 (23.15)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.0873, Mixed Models Analysis; Mean Difference (Net) = -12.6627, 95% CI 2-sided [-27.2243 to 1.8989], Standard Error of Mean 7.3097
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.2866, Mixed Models Analysis; Mean Difference (Net) = -7.3578, 95% CI 2-sided [-21.0154 to 6.2999], Standard Error of Mean 6.8559

7. Other Pre Specified Outcome: PCL-5 (Post-Traumatic Stress Disorder Checklist)
Description: The PCL is a validated 20-item, self-report measure of PTSD symptoms. Items are rated from 0 to 4 (0 = not at all, 4 = extremely). Total scores range from 0-80. Higher scores indicate higher post-traumatic stress symptoms.
Time Frame: Baseline
Population: This measure was only collected at baseline. The number analyzed in one or more rows differs from overall number analyzed because some participants chose to not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 24 | 24
score on a scale | 33.29 (17.62) | 29.25 (20.67)

8. Other Pre Specified Outcome: Patient Health Questionnaire - PHQ-9
Description: The PHQ-9 is a reliable and well-validated self-report measure of depressive symptom severity and suicide risk based on Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria. Items are rated from 0 to 3 (0 = not at all, 3 = nearly every day). Total scores range from 0 to 27. Totals are categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), and severe (20-27).
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 22 | 23
score on a scale
  3 months | 9.27 (6.28) | 10.83 (5.11)
  6 months: number analyzed (Participants) | 18 | 16
  6 months | 8.61 (5.46) | 7.88 (4.88)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.2776, Mixed Models Analysis; Mean Difference (Net) = -1.5655, 95% CI 2-sided [-4.4168 to 1.2859], Standard Error of Mean 1.4313
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.6636, Mixed Models Analysis; Mean Difference (Net) = 0.7202, 95% CI 2-sided [-2.5651 to 4.0055], Standard Error of Mean 1.6492

9. Other Pre Specified Outcome: Generalized Anxiety Disorder (GAD-7)
Description: The GAD-7 is a reliable and validated 7-item, self-report measure of anxiety. Items are rated from 0 to 3 (0 = not at all, 3 = nearly every day). Total scores range from 0 to 21 and are categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), and severe (15-21) anxious symptoms.
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 23 | 21
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 9.04 (6.43) | 6.78 (4.17)
  6 months | 8.30 (6.28) | 8.90 (4.99)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.1733, Mixed Models Analysis; Mean Difference (Net) = 2.3254, 95% CI 2-sided [-1.0443 to 5.695], Standard Error of Mean 1.6911
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.7398, Mixed Models Analysis; Mean Difference (Net) = -0.5408, 95% CI 2-sided [-3.7726 to 2.6911], Standard Error of Mean 1.622

10. Other Pre Specified Outcome: Veterans RAND 12 (VR-12)
Description: The VR-12 is a 12-item measure used to assess health related quality of life and to produce physical and mental health component scores. The 12 items are summed into a physical component score (PCS) and a mental component score (MCS). Both the PCS and MCS scores are transformed to a scale with a range of 1-100. A higher score indicates better health.
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 23 | 22
score on a scale
  Physical Component Scale - 3 months: number analyzed (Participants) | 23 | 18
  Physical Component Scale - 3 months | 41.84 (5.14) | 41.94 (4.15)
  Physical Component Scale - 6 months | 39.93 (5.90) | 40.20 (4.85)
  Mental Component Scale - 3 months: number analyzed (Participants) | 23 | 18
  Mental Component Scale - 3 months | 34.56 (10.15) | 34.81 (5.95)
  Mental Component Scale - 6 months | 35.02 (7.78) | 38.02 (6.15)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; Physical Component Scale - 3 months; Test type: Superiority; p = 0.9239, Mixed Models Analysis; Mean Difference (Net) = -0.1491, 95% CI 2-sided [-3.2476 to 2.9494], Standard Error of Mean 1.5551
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; Physical Component Scale - 6 months; Test type: Superiority; p = 0.8456, Mixed Models Analysis; Mean Difference (Net) = -0.2879, 95% CI 2-sided [-3.2238 to 2.6481], Standard Error of Mean 1.4735
Statistical Analysis 3: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; Mental Component Scale - 3 months; Test type: Superiority; p = 0.9413, Mixed Models Analysis; Mean Difference (Net) = -0.1757, 95% CI 2-sided [-4.9175 to 4.5661], Standard Error of Mean 2.3798
Statistical Analysis 4: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; Mental Component Scale - 6 months; Test type: Superiority; p = 0.1934, Mixed Models Analysis; Mean Difference (Net) = -2.9597, 95% CI 2-sided [-7.4526 to 1.5333], Standard Error of Mean 2.2549

11. Other Pre Specified Outcome: Insomnia Severity Index (ISI)
Description: The ISI is a 7-item measure of the participant's perceptions of their insomnia, such as severity of sleep-onset and sleep maintenance difficulties. Items are rated from 0 to 4 (0 = not at all, 4 = very much). Total scores range from 0 to 28. Totals are categorized as follows: no clinically significant insomnia (0-7), subthreshold insomnia (8-14), clinical insomnia (moderately severe) (15-21), clinical insomnia (severe) (22-28).
Time Frame: 3 and 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 23 | 21
score on a scale
  3 months: number analyzed (Participants) | 23 | 18
  3 months | 16.35 (7.44) | 13.28 (6.45)
  6 months: number analyzed (Participants) | 22 | 21
  6 months | 16.91 (8.74) | 14.86 (5.48)
Statistical Analysis 1: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 3 months; Test type: Superiority; p = 0.1442, Mixed Models Analysis; Mean Difference (Net) = 3.0999, 95% CI 2-sided [-1.0852 to 7.2849], Standard Error of Mean 2.1004
Statistical Analysis 2: Comparison: TENACITY Telehealth Cognitive Behavioral Therapy for Migraine vs Behavioral Usual Care; 6 months; Test type: Superiority; p = 0.3132, Mixed Models Analysis; Mean Difference (Net) = 2.0675, 95% CI 2-sided [-1.9892 to 6.1243], Standard Error of Mean 2.036

12. Primary Outcome: Budget Impact Analysis - Time
Description: Time associated with program implementation
Time Frame: 2 years
Population: Summary Time (hours of training)
Measure: Number; unit: hours
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 30 | 27
hours | 201.1 | 4.0

13. Primary Outcome: Budget Impact Analysis - Cost Per Veteran
Description: Costs associated with intervention per Veteran
Time Frame: 2 years
Population: Summary Costs
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
Number analyzed (Participants) | 30 | 27
dollars | 194.46 (107.47) | 113.52 (210.40)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 7 months after participants started treatment which was the end of the study period.
Description: Adverse event collection was performed by participant self-reporting to study personnel.
Arm/Group | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine | Behavioral Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/27
Serious Adverse Events (participants affected / at risk) | 1/30 | 3/27
Other Adverse Events (participants affected / at risk) | 13/30 | 10/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine (N=30) | Behavioral Usual Care (N=27)
colitis (Gastrointestinal disorders) | 1 | 0
stomach pain (Gastrointestinal disorders) | 0 | 1
bowel obstruction (Gastrointestinal disorders) | 0 | 1
flu (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TENACITY Telehealth Cognitive Behavioral Therapy for Migraine (N=30) | Behavioral Usual Care (N=27)
allergic reaction (Immune system disorders) | 0 | 1
arm/leg pain (Musculoskeletal and connective tissue disorders) | 1 | 0
arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
chest pain (Cardiac disorders) | 0 | 1
GERD (Gastrointestinal disorders) | 1 | 0
COVID (Infections and infestations) | 0 | 3
dehydration (General disorders) | 0 | 1
depressive symptoms (Psychiatric disorders) | 2 (3) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 | 0
fall (Injury, poisoning and procedural complications) | 2 (3) | 0
fever (Infections and infestations) | 1 | 0
flu (Infections and infestations) | 2 | 0
foot pain (Metabolism and nutrition disorders) | 1 | 0
hernia (Gastrointestinal disorders) | 0 | 1
hives (Immune system disorders) | 0 | 1
insomnia (General disorders) | 0 | 1
irregular heartbeat (Cardiac disorders) | 1 | 0
leg pain (Musculoskeletal and connective tissue disorders) | 1 | 1
migraine (General disorders) | 1 (2) | 0
pain symptoms (Musculoskeletal and connective tissue disorders) | 1 | 2
plantar wart (Skin and subcutaneous tissue disorders) | 1 | 0
PTSD (Psychiatric disorders) | 0 | 1
rash (Skin and subcutaneous tissue disorders) | 0 | 1
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1
sinus infection (Infections and infestations) | 1 | 0
stomach virus (Infections and infestations) | 0 | 1
superficial burn (Injury, poisoning and procedural complications) | 1 | 0

LIMITATIONS AND CAVEATS:
Limitations include not reaching the target number of participants needed to achieve sufficient statistical power. We initially consented 80 participants of which 57 of the 80 were eligible to be randomized based on the 30 day headache diary outcomes confirming chronic headache. The study was conducted during the COVID-19 pandemic. Thus, the enhanced headache usual treatment was often offered via telehealth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/62/NCT04613362/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04613362/ICF_000.pdf